CLINICAL TRIAL: NCT00574574
Title: Biological Effects of an Anthocyanin Rich Dietary Supplement on Skin Ageing and Markers of Inflammation in Post-Menopausal Women
Brief Title: Effects of Anthocyanin on Skin Health and Markers of Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other); Unilever R&D (Industry)
Responsible Party: Prof Aedin Cassidy, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R14764; BWF008
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Cardiovascular Disease; Skin Health; Postmenopause
Keywords: cardiovascular disease; CVD; skin health; postmenopausal women; anthocyanin; inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 500mg/d of anthocyanin, contained in 4 X 250mg capsules (125mg anthocyanin/ capsule). 2 capsules to be taken with food, twice per day (n=4 in total).
  Interventions: Dietary Supplement: anthocyanin
- 2 (Placebo Comparator): 500mg/d of placebo control containing no anthocyanin, 2 X 250mg capsules to be taken with food, twice per day (n=4, 250mg capsules in total / d).
  Interventions: Dietary Supplement: anthocyanin

INTERVENTIONS:
Dietary Supplement: anthocyanin — 500mg/d of anthocyanin each day for 12 weeks (84days). Route of administration: oral capsules, 4 X 250mg capsules (125mg anthocyanin/ capsule). Dosage advice; 2 capsules to be taken with food, twice per day (n=4 in total).

SUMMARY:
The purpose of this study is to determine whether short-term exposure to a compound found in some fruits and vegetables (anthocyanin), is effective in improving skin health and reducing the levels of various markers of cardiovascular disease risk. A range of skin health parameters are being studied and volunteers are also providing skin biopsy, urine and blood samples. 62 postmenopausal women have been recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Upper age limit of 70 years
* Minimum of 1 year since last menstruation
* Not taking Hormone Replacement Therapy (HRT), and not having taken HRT for a minimum of 6 months prior to commencement
* Having no significant past or present medical history of: inflammatory conditions (including eczema, asthma, hay fever, IBS, crohn's disease and arthritis), diabetes, hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, thyroidal or psychiatric disease.
* Agreeing to restrict dietary intake of anthocyanin containing foodstuffs and also other foodstuffs considered to be cardio-protective i.e. red wine, total alcohol, oily fish, dark chocolate, tea and coffee.
* Agreeing to maintain existing cosmetic and beauty regime, and avoid 'tanning' (either naturally or synthetically) of the specific sites of skin function measurement during the study.
* BMI 20-32 kg/m2
* Successful biochemical, haematological and urinalysis assessment

Exclusion Criteria:

* allergy / sensitivity to local anaesthetic i.e. Xylocaïne
* Regular use of aspirin, or other anti-inflammatory pain relief medication, as prescribed by a doctor. [If subjects are regular self prescribed aspirin users and are willing to give up aspirin 2 months prior to the study and for the duration of the study they can be included.]
* Taking other counter indicative medication e.g. steroidal medication during the trial, or within 1 month of the trial beginning.
* Taking food / dietary supplements e.g. vitamins, minerals, fish oils, plant oils, isoflavones, soy products, carotenoids during the trial (unless prepared to cease intake during, and 1 month preceding the trial).
* Those on therapeutic diets or following weight-loss diet.
* Current smoker, or smoker in the past year
* Having vaccinations or antibiotics within 3 months of start of trial, and those with vaccinations scheduled for during the trial
* Parallel participation in another research project which involves dietary intervention and/or sampling of biological fluids/material
* Participation in another research project within the last four months unless the total amount of combined blood from both studies will not exceed 470ml.
* Those intending to travel during the study to locations where a change in skin colour may be anticipated
* Subjects intending to deliberately "sunbathe", use tanning solariums or tanning creams on body sites used for assessment.
* Assessed from the clinical screening
* abnormal renal function (Na >145mmol/L, K >5.0mmol/L, Urea >7.1mmol/L, Albumin >50g/L, Creatinine >125μmol/L, Total bilirubin >22μmol/L), or liver function (ALP >126 IU/L, ALT >50 IU/L), lipid profile (Total cholesterol > 6.5 mmol/l, TAG >3.0 mmol/l, HDL>2.0 mmol/l), anaemia (Haemoglobin <11.5g/dL), fasting glucose (> 6.1 mmol/l) or measurements considered to be counter indicative of the trial outcome measures.
* Untreated hypertension (>160/90mmHg) or hypotension (90/50mmHg or 95/50mmHg if symptomatic)
* BMI <19.5 or >32.5

Max Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Measure: Evidence of significant differences in skin health parameters, between active treatment and placebo supplementation period. | 12 Weeks

SECONDARY OUTCOMES:
Measure: Evidence of significant differences in inflammatory status, between active treatment and placebo supplementation period. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aedin MM Cassidy, PhD, Principal Investigator — UEA
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom